CLINICAL TRIAL: NCT06237257
Title: A Study of Chemoradiotherapy With SHR-1316 For Treatment of Locally Advanced Cervical Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-202
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-04

CONDITIONS: Locally Advanced Cervical Cancer
MeSH Terms: interventions — Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1316 plus concurrent chemoradiotherapy (Experimental)
  Interventions: Biological: SHR-1316; Drug: Cisplatin Injection/Carboplatin Injection; Radiation: External Beam Radiotherapy (EBRT)/Brachytherapy; Drug: Paclitaxel Injection

INTERVENTIONS:
Biological: SHR-1316 — SHR-1316（Adebrelimab Injection）
Drug: Cisplatin Injection/Carboplatin Injection — Cisplatin Injection/Carboplatin Injection
Radiation: External Beam Radiotherapy (EBRT)/Brachytherapy — External Beam Radiotherapy (EBRT)/Brachytherapy
Drug: Paclitaxel Injection — Paclitaxel Injection.

SUMMARY:
The Primary purpose of this study is to evaluate the safety of SHR-1316 plus concurrent chemoradiotherapy in participants with locally advanced cervical cancer.

The second purpose of this study is to evaluate the efficacy and PK traits; The exploratory study is to explore the biomarker 、immunogenicity and so on .

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Has histologically-confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix；
3. Has locally advanced cervical cancer；
4. At least one measurable lesion ( RECIST version 1.1)；
5. Investigator assess it is suitable for concurrent chemoradiotherapy;
6. Has provided a tissue sample from tumor lesion;
7. Cooperative Oncology Group (ECOG) performance status of 0 or 1;
8. BMI≥18.5kg/m2；
9. Female participants of childbearing potential must agree to use highly effective contraception during the treatment period and for at least 7 months after the last dose of drug，Female participants' HCG must be negative within 3 days prior to enrollment and must be non-lactating.

Exclusion Criteria:

1. Histopathologically confirmed small cell carcinoma (neuroendocrine) or mucinous adenocarcinoma of the cervix；
2. The presence of distant metastatic disease was confirmed by pathology or imaging;
3. has previously undergone hysterectomy (including subtotal hysterectomy) or plan to undergo hysterectomy for cervical cancer, or plan to adopt fertility preservation therapy;
4. In the investigator's judgment, there is a disease (such as severe diabetes, neurological or psychiatric illness, etc.) or any other condition that seriously endangers the subject's safety, confuses the study results, or interferes with the subject's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Type, incidence and grade of drug-related adverse events of grade 3 and above | Up to approximately 24 months

SECONDARY OUTCOMES:
Adverse events (AEs) include incidence, grade (judged according to NCI-CTCAE V5.0 standards), duration and correlation with study drugs | Up to approximately 30 months
Rate of Suspension and Discontinuation Due to an Adverse Event correlation with study drug | Up to approximately 30 months
Objective Response Rate(ORR) | Up to approximately 60 months
  judged based on RECIST 1.1 criteria according to Investigator's assessment
Duration of response (DoR) | Up to approximately 60 months
  judged based on RECIST 1.1 criteria according to Investigator's assessment
Progression free survival (PFS) | Up to approximately 60 months
  judged based on RECIST 1.1 criteria according to Investigator's assessment
Overall Survival (OS) | Up to approximately 60 months
  judged based on RECIST 1.1 criteria according to Investigator's assessment
2-year Progression free survival | Up to approximately 24 months
  judged based on RECIST 1.1 criteria according to Investigator's assessment
3-year Overall Survival | Up to approximately 36 months
  judged based on RECIST 1.1 criteria according to Investigator's assessment
12-week Complete Response | Up to approximately 4 months
  judged based on RECIST 1.1 criteria according to Investigator's assessment
PK traits of SHR-1316: Cmax | Up to approximately 24 months
PK traits of SHR-1316: Tmax | Up to approximately 24 months
PK traits of SHR-1316: AUC0-t | Up to approximately 24 months
PK traits of SHR-1316: AUC0-∞ | Up to approximately 24 months
PK traits of SHR-1316: t1/2 | Up to approximately 24 months
PK traits of SHR-1316: CL | Up to approximately 24 months
PK traits of SHR-1316: Vss | Up to approximately 24 months
Serum concentration of SHR-1316 at each planned blood collection time point | Up to approximately 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided